CLINICAL TRIAL: NCT06332131
Title: Effects of Immune Checkpoint Inhibitors on Coronary Microvasculature
Status: Enrolling by invitation | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC07623
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Coronary Microvascular Dysfunction; Cardiotoxicity; Breast Cancer; Lung Cancer (NSCLC)
Keywords: cancer therapy related cardiotoxicity; Immune checkpoint inhibitor therapy
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be collected and banked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study that includes patients with breast cancer or non-small cell lung cancer who will be treated with immune checkpoint inhibitor (ICI) therapy. The investigators will use echocardiograms, blood draws, and PET stress tests to understand how ICI therapy affects the heart and circulatory system.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Either diagnosis of breast cancer with plan for treatment according to the Keynote 522 regimen or non-small-cell lung cancer planned for neoadjuvant treatment that includes pembrolizumab
* Able to provide written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding:
* Prior treatment with ICI therapy.
* Vulnerable patients, including pregnant women and prisoners
* Absolute Contraindication to rest/vasodilator stress PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast or lung cancer planned for treatment that includes pembrolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of new abnormal myocardial blood flow reserve (MBFR) | 3 months
  Development of MBFR<2

SECONDARY OUTCOMES:
Incidence of major cardiovascular events | 3 months
  Composite measure including new/worsened heart failure, MI, stroke, myocarditis
Coronary calcium score | 3 month
  Change in PET derived Coronary Calcium (CAC) Score from baseline. CAC ranges from 0-400 agatson units; higher CAC indicates larger amounts of calcium are present in the coronary arteries.
All cause mortality | 3 months
  All cause mortality
Cardiovascular specific mortality | 3 months
  Cardiovascular specific mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Scherrer-Crosbie, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided